CLINICAL TRIAL: NCT04438564
Title: Immunoassay and Regulation of Traditional Chinese Medicine on Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH108-REC1-113
Record Dates: First submitted 2020-06-14; First posted 2020-06-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Cancer of Ovary; Cancer of Endometrium
Keywords: Chinese Herbal Medicine, Immunity, T Cell, Dendritic Cell
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cancer of breast, colorectal, ovarian and endometrial (Other): Patient who diagnostic of Breast cancer, Colorectal cancer, cancer of Ovary, and cancer of Endometrial are can recruit.
  Interventions: Other: Cases for patients diagnosed with breast cancer, colonrectal cancer, ovarian cancer and endometrial cancer

INTERVENTIONS:
Other: Cases for patients diagnosed with breast cancer, colonrectal cancer, ovarian cancer and endometrial cancer — Diagnosis and acceptance of breast cancer, colon rectal cancer, ovarian cancer, and endometrial cancer by the clinical Western medicine team.

SUMMARY:
The immune system is our body's defense mechanism, which helps us to resist foreign pathogens and cancer cells in the body. However, if the immune system is too weak, too strong, or unbalanced, it will be susceptible to get bacterial and viral infections, unable to fight cancer, or cause allergies, autoimmune and rheumatic diseases. At present, there is no good western medicine to strengthen immunity when the body is insufficient immunity. However, strong immunity causes autoimmune diseases and need to be treated by steroids and immunosuppressive agents. These drugs have limited efficacy and often have many side effects. In the clinical practice of traditional Chinese medicine, tonify qi, supplement blood and nourish yin are often used to enhance immunity. However, there is no clinical test to demonstrate the modulation of immune response after traditional Chinese medicine treatment.

In our preliminary study, the investigators identified that the basic immune response of cancer patients is weaker than healthy people by testing the level of IFN-r (promoting T cell activity, anti-tumor, anti-viral), TNF-a (promoting B cell proliferation, producing antibodies, anti-tumor, anti-viral) and IL-2 (regulate the proliferation and differentiation). Besides, some Chinese herbal extracts can significantly stimulate the immune response higher than the general average basic immunity of cancer patients. Further, we will use the stimulatory Chinese medicine extract to administer to cancer patients and examine the immune response of cancer patients after taking them. Therefore, this test can provide actual data on the basic immunity of healthy people or cancer patients and the modulation of immune response by traditional Chinese medicine treatment. This analysis platform provides patients to select the medicines that can enhance the immune response for individuals and analyze the changes of the immune response after conditioning with the candidate Chinese medicines. Therefore, this test could be applied clinically to validate the immunological regulation of Chinese herbal medicine as well as analyze the immunological modulation against different cancer by various Chinese herbal medicine.

DETAILED DESCRIPTION:
Traditional Chinese medicine (TCM) and dendritic cells (DCs) activation/maturation One of the important approaches to successful cancer immunotherapy is generation of specific T cell responses by dendritic cells (DCs). DCs are the most potent antigen-presenting cells for naive T cells, because their high expression of MHC and co-stimulatory molecules. DCs comprise several subsets, and their roles in the presentation of antigens derived from pathogens, vaccines and self tissues are now beginning to be elucidated. Immature DCs (iDCs) resided in periphery have a high ability to endocytose antigens and become to mature DCs (mDCs) upon a variety of stimuli through Toll-like receptors (TLRs). However, iDCs facilitate immune tolerance and fully mDCs can promote immune responses. Until now, there are some studies have demonstrated that TCM could promote the activation status of DC to enhance immune responses through TLR, which are characterized by increased expression of co-stimulatory moleculars, MHC class II and several cytokines. Ganoderma lucidum and Cordyceps sinensis have been widely used in Asian countries to have beneficial effects on human health. Ganoderma lucidum polysaccharides have been reported to induce DCs maturation and promote the cytotoxicity of specific CTL. Moreover, Ganoderma lucidum polysaccharides were able to induce DC activation markers production and cytokines expression through TLR-4 signaling pathway. However, this character about TCM acted as TLR agonists could apply to develop safe and effective adjuvant in vaccine generation.

Traditional Chinese medicine (TCM) and T cell activation T cells are the master regulators of adaptive immune responses. Proper T cell responses are essential for the hosts to orchestrate sufficient adaptive immunity. Classically, the TH1/TH2 hypothesis has served the immunology community well, particularly in understanding infectious and allergic diseases. Regulatory T cells (Treg) are suppressive T cells that regulate effector T cell immunity. Nevertheless, this model dose not fit all systems when it comes to the study of organ-specific autoimmune diseases. It has also become more and more clear, however, that many complicated pathological situations cannot be simply explained by the TH1 cell and TH2 cell paradigm. Efforts to resolve these issues in recent years have resulted in the discovery of TH17 cells.

T cell immunity is crucial for anti-tumor immunity. Given their importance in immune responses and diseases, it is important to understand the regulation of T cell immunity. In immune system, different lineages of immune cells were conventionally distinguished by the morphology and expression of a cluster of differentiation markers on the cell surface. TH1 cells that make IL-2 and IFN-r are important for delayed-type hypersensitivity reactions, whereas TH2 cells that make IL-4 promote IgE production and allergic reaction. The differentiation of TH1 and TH2 cells mainly through the induction of distinct transcriptional programs. Activation of Signal Transducers and Activators of Transcription 1 (STAT1) by IFN-r and STAT4 by IL-12 drives expression of T-bet for TH1 programming. On the other hand, activation of STAT6 by IL-4 promotes GATA3 expression in TH2 cells. A revise of the TH1/TH2 hypothesis was proposed until the discovery and IL-23 and IL-17. TH17 cell is a distinct T helper cell population that plays a crucial role in CD4+ T cell-mediated adaptive immunity. Commitment to the TH17 pathway requires the presence of both IL-6 and TGF-a during in vitro culture. These cells, different from the classical TH1 and TH2 cells, do not produce IFN-r or IL-4 but on the other hand express the IL-23 receptor and IL-21, IL-22, and IL-17F. ROR-rt , ROR-rt are also highly expressed in TH17cells and can be induced by TGF-a and IL-6. Our previous studies showed for the first time an in vivo requirement for STAT3 in TH17 mediated autoimmunity. In addition, the investigators found that STAT3 is required for the maintenance of endogenous TH17 cells. In a more recent report, the investigators also found that CD8 T cells, like their CD4 counterparts TH17, can be skewed toward IL-17 production in vitro and in vitro.

Manipulating T cell immunity by Chinese herbs is a promising field to explore. Many herbs were reported to regulate the T cell activation. Tanshinlactone A from Salvia miltiorrhiza Bunge significantly decreased the IL-2 and IFN-γ gene expression through reduction of MAPK activation in phytohemagglutinin-activated peripheral blood mononuclear cells. Periplocoside E (PSE) was shown to dose-dependently inhibit anti-CD3 induced primary T cell proliferation, activation for IL-2R (CD25) expression, and IFN-γ and IL-2 production at the transcriptional level by inhibited the activation of ERK and JNK. Furthermore, kurarinol was reported to increase level of HBV specific CTL by down-regulating peripheral blood HBV specific CTL surface PD-1 expression of CHB patients.

All of these will support investigators' hypothesis that modulation of dendritic cell and T cell immunity by Chinese herbs or cytokines may be an applicable intervention to modulate immunity, for example, to promote anti-tumor immunity against cancer. The successful completion of the proposed studies will provide a strong support for future development of anti-cancer immunotherapy by Chinese herbs.

Traditional Chinese herbs as a pharmacologic approach to modulate immunity Cancer immunotherapy, allergy, and autoimmune diseases are among the chronic illness that accounts for the death and economic burdens in Taiwan and other modern countries. Diseases such of Rheumatoid arthritis (RA), SLE, multiple sclerosis, ankylosing spondylitis, vasculitis, psoriasis and Sjogren's syndrome are common autoimmune diseases that cause not only life-long discomfort but also disabilities of the patients. Cancer immunotherapy is promising. Many of autoimmune disease and difficult-to-treat allergies are now found to be associated with IL-17 mediated pathology. However, the current treatment is limited. Recently, targeted therapy such as Etanercept (trade name Enbrel), a biopharmaceutical that interferes with tumor necrosis factor (TNF; a soluble inflammatory cytokine), has been developed to treat some of the autoimmune diseases. However, nhibition of TNF has substantially advanced the treatment of inflammatory diseases. Because TNF and IL-17 have shared functions, the rationale for testing IL-17 inhibitors in the clinic is often based on the concept that patients who do not respond to TNF inhibitors may have an IL-17-driven disease. Autoimmune diseases such of rheumatoid arthritis and multiple sclerosis are common autoimmune diseases that cause not only life-long discomfort but also disabilities of the patients. The current treatment for these autoimmune diseases is limited to analgesia, anti-inflammatory drugs, steroids, disease-modifying antirheumatic drugs (DMARDs), and immunosuppressants. Recent studies in mouse models and in humans have identified a key role of IL-17 and TH17 cells in the pathogenesis of inflammation and autoimmunity as well as in host defense against certain pathogens.

Meanwhile, there are some studies using Chinese herbs to modulate CD4 TH17 immunity. Compound extracted from Chinese herbs, such as berberine exhibited potent efficacy inhibiting TH17 in the EAE model. Triptolide also inhibited collagen-induced arthritis (CIA), a model of rheumatoid arthritis, through inhibition of CD4 TH17 cells. Periplocoside A was found to ameliorate EAE by suppressing IL-17 production and inhibited the differentiation of Th17 cells in vitro. Eriocalyxin B was also found to be effective to inhibit TH17 and EAE through targeting Janus Kinase/Signal Transducer and Activator Of Transcription and Nuclear factor-kappaB signaling pathways. TCM formula such as Qingkailing injection was found to ameliorate rat experimental autoimmune uveitis (EAU). Qingkailing injection can alleviate autoimmune uveitis in rats, inhibit the differentiation toward Th1 and Th17 effector cells and the relevant cytokines secretion. Pure compound from Daphne odora var. marginata (D. marginata) was also found to inhibit TH17 and thus exhibit inhibitory effects in CIA model.

One of the landmark study published in Science and Nature Chemical Biology is the example of halofuginone, an active component of traditional Chinese herb hydrangea root (Dichroa febrifuga), used to treat malaria for thousands of years. A collaborative research team led by Dr. Mark Sundrud at the Department of Pathology, Harvard Medical School and Immune Disease Institute, Boston, MA, has reported that halofuginone halted the progression of experimental autoimmune encephalomyelitis (EAE) mice and TH17. Importantly, unlike other therapies for autoimmune diseases, halofuginone does not have the undesirable effect of suppressing the other immune system.

The investigators have established some platforms for screening Chinese herbs not only for modulating PD-1/PD-L1, IL-17, but also for detection of dendritic cell and T cell activation (Immunogen Test Panel).

The hypothesis is that modulation of dendritic cells and T cells by traditional Chinese medicine may be an applicable intervention to treat some of the immunologic diseases such as cancer, allergy, and autoimmune diseases. Studies that can fit the niche, understanding the function and mechanism of Chinese herbs on immune cells and its pathway, will have broad clinical and immunological significance. The successful completion of the proposed studies will provide a strong support for a clinical trial of traditional Chinese medicine to treat patients with immunologic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ovarian cancer and endometrial cancer (cancer patients treated with chemotherapy, radiotherapy, and surgery) can be included.
* Breast cancer: Diagnosed by pathological diagnosis of biopsy, without chemotherapy or radiotherapy.
* Colorectal cancer: Diagnosed by pathological diagnosis of slices, without chemotherapy or radiotherapy.

Exclusion Criteria:

* Pregnant women
* Minors under the age of 20.
* Those who are currently using traditional Chinese medicine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The IL-2, TNF-alpha and IFN-gamma expression by traditional Chinese medicine treatment on cancer patients | one year
  The cytokines expression of immune cells in the blood by traditional Chinese medicine treatment in breast cancer, colon-rectal cancer, ovarian cancer, and endometrial cancer will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: China Medicine University, Study Chair — China Medicine University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan